CLINICAL TRIAL: NCT06824493
Title: Orthodontic Treatment on Oral Microbiota and Salivary Proteins
Status: Not yet recruiting | Type: Observational
Sponsor: Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Shanshan-Dai, attending physician of pediatric dentist and PhD in Orthodontics, Xi'an Jiaotong University
Other Study IDs: XJKQLY202503
Record Dates: First submitted 2025-01-11; First posted 2025-02-13 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Orthodontics; White Spot Lesions [Initial Caries] on Smooth Surface of Tooth; Caries, Dental
Keywords: microbiota
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ID number
  Interventions: Other: no interventions; Other: None-placebo; Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: no interventions — no intervention as this is an observational studies
Other: None-placebo — Observational study with no interventions
Other: No Intervention: Observational Cohort — no intervention because of observational studies

SUMMARY:
Study on the changes in oral microbiota during orthodontic treatment in patients aged 8-18 years. Orthodontic patients treated at Stomatology Hospital of Xi'an Jiaotong University from March 2025 to March 2027 will be recruited. Prior to orthodontic treatment, routine preoperative examinations will be conducted, informed consent forms will be signed, baseline oral conditions will be recorded, and oral and psychological-related questionnaires will be completed. Patients will be informed of the need for regular oral hygiene check-ups, caries risk assessments will be performed, and plaque, saliva, and intraoral photographs will be collected. During orthodontic treatment, plaque samples will be collected every 3 months, and saliva samples will be collected every 6 months until the treatment is completed to evaluate the changes in oral microbiota throughout the orthodontic process.

ELIGIBILITY:
Inclusion Criteria:

* No carries and White spot
* No missing teeth
* No history of oral treatment
* No malocclusion
* No systemic diseases

Exclusion Criteria:

* Antibiotic use in the past three months
* A history of long-term medication use
* A history of dental fillings
* Unable to attend regular follow-ups

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A description of the population from the population undergoing oral health examinations in primary schools
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Microbiota changes of plaque | baseline, collect plaque in the first month, then at Month 3, 6, 9, 12, 15, 18, 21, 24, 27,30 through study completion, an average of 30 months.
  Samples of supragingival plaques will proceed to 16S rRNA sequencing for analysis of microbiome profiles, and q-PCR for evaluating bacterial loads of some critical pathogens for dental caries
Microbiota changes of saliva | Baseline, collect saliva at Months 6, 12, 18, 24, 30 through study completion, an average of 30 months.
  Samples of saliva will proceed to 16S rRNA sequencing for analysis of microbiome profiles, and q-PCR for evaluating bacterial loads of some critical pathogens for dental caries
Monitoring dental lesion progression | Baseline, follow-up assessments are conducted at Months 6, 12, 18, 24, 30 through study completion, an average of 30 months.
  ICDAS(International Caries Detection and Assessment System) scoring system helps in detecting early caries, monitoring lesion progression, and developing tailored treatment strategies. Scoring Criteria: 0: No visible caries; 1: First visual change (only visible when dry); 2: Distinct visual change (visible without drying); 3: Initial enamel breakdown;4: Underlying dark shadow from dentin;5: Moderate cavity with dentin exposure; 6: Extensive cavity with pulp involvement